CLINICAL TRIAL: NCT00260286
Title: Dietary Energy Requirements in Physically Active Men and Women, Objective 4B: Effects of Gynecological Age on LH Sensitivity to Energy Availability
Brief Title: Effects of Gynecological Age on LH Sensitivity to Energy Availability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio University (Other)
Collaborators: Ohio State University (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: Excalibur X; DAMD_17-95-1-5053,; M01RR000034 (NIH)
Record Dates: First submitted 2005-11-30; First posted 2005-12-01 (Estimated); Last update posted 2005-12-05 (Estimated); Status verified 2005-11

CONDITIONS: Anovulation; Amenorrhea; Infertility; Starvation
Keywords: LH pulsatility; energy availability; exercise; diet; gynecological age
MeSH Terms: conditions — Anovulation; Amenorrhea; Infertility; Starvation; Motor Activity

INTERVENTIONS:
Behavioral: Energy availability

SUMMARY:
The purpose of this experiment is to investigate whether the dependence of luteinizing hormone pulsatility on energy availability declines during adolescence.

DETAILED DESCRIPTION:
The incidence of menstrual disorders declines during adolescence. This has long been attributed to the gradual "maturation" of the hypothalamic-pituitary-ovarian axis, but the mechanism of this "maturation" is not known. Ovarian function critically depends on the pulsatile secretion of gonadotropin-releasing hormone (GnRH) by the hypothalamus and on the consequent and more readily assessed pulsatility of luteinizing hormone (LH) secretion by the pituitary. LH pulsatility has been shown to depend on energy availability, operationally defined as dietary energy intake minus exercise energy expenditure. The effects of energy availability on LH pulsatility are thought to be mediated by certain metabolic substrates and hormones.

Comparison: By manipulating diet and exercise regimens, contrasting energy availability treatments of 10 and 45 kilocalories per kilogram of fat-free mass per day are being administered to adolescents with 5-8 years of gynecological age and to adults with 14-18 years of gynecological age for five days in the early follicular phase of separate menstrual cycles. Effects of low energy availability on LH pulsatility and on selected metabolic substrates and hormones are being measured.

ELIGIBILITY:
Inclusion Criteria:

* 5-8 or 14-18 years of gynecological age
* menstrual cycles of 26 to 32 days for the previous 3 months
* luteal phase length >11 days
* 18-32% body fat

Exclusion Criteria:

* smoking
* oral contraceptives
* hematocrit <35%
* diet with <35 or >55 kcal/kgFFM/day of energy
* habitually performing more than 60 minutes/week of aerobic exercise
* histories or evidence of heart, liver, or kidney disease, diabetes, menstrual or thyroid disorders, pregnancy, lactation, and congenital or acquired orthopedic abnormalities

Ages: 18 Years to 34 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18
Dates: Start 2001-08; Study Completion 2004-05

PRIMARY OUTCOMES:
Differences in 24h LH pulse frequency, 24h LH pulse amplitude and 24h LH mean concentration in blood samples drawn q10' for 24 hours after 5 days of treatment

SECONDARY OUTCOMES:
Differences in 24h average glucose, beta-hydroxybutyrate, insulin, cortisol, growth hormone, insulin-like growth factor-I, tri-iodothyronine, and leptin concentrations in blood samples drawn q10' for 24 hours after 5 days of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Anne B Loucks, Ph.D., Principal Investigator — Ohio University
Locations (1):
- Ohio University, Athens, Ohio, United States

REFERENCES:
- [Background] Loucks AB, Verdun M, Heath EM. Low energy availability, not stress of exercise, alters LH pulsatility in exercising women. J Appl Physiol (1985). 1998 Jan;84(1):37-46. doi: 10.1152/jappl.1998.84.1.37. PMID 9451615
- [Background] Loucks AB, Heath EM. Induction of low-T3 syndrome in exercising women occurs at a threshold of energy availability. Am J Physiol. 1994 Mar;266(3 Pt 2):R817-23. doi: 10.1152/ajpregu.1994.266.3.R817. PMID 8160876
- [Background] Hilton LK, Loucks AB. Low energy availability, not exercise stress, suppresses the diurnal rhythm of leptin in healthy young women. Am J Physiol Endocrinol Metab. 2000 Jan;278(1):E43-9. doi: 10.1152/ajpendo.2000.278.1.E43. PMID 10644535
- [Background] Loucks AB, Callister R. Induction and prevention of low-T3 syndrome in exercising women. Am J Physiol. 1993 May;264(5 Pt 2):R924-30. doi: 10.1152/ajpregu.1993.264.5.R924. PMID 8498602
- [Background] Loucks AB, Heath EM. Dietary restriction reduces luteinizing hormone (LH) pulse frequency during waking hours and increases LH pulse amplitude during sleep in young menstruating women. J Clin Endocrinol Metab. 1994 Apr;78(4):910-5. doi: 10.1210/jcem.78.4.8157720.
- [Background] Loucks AB, Verdun M. Slow restoration of LH pulsatility by refeeding in energetically disrupted women. Am J Physiol. 1998 Oct;275(4):R1218-26. doi: 10.1152/ajpregu.1998.275.4.R1218. PMID 9756553
- [Background] Loucks AB, Thuma JR. Luteinizing hormone pulsatility is disrupted at a threshold of energy availability in regularly menstruating women. J Clin Endocrinol Metab. 2003 Jan;88(1):297-311. doi: 10.1210/jc.2002-020369. PMID 12519869
- [Background] Ihle R, Loucks AB. Dose-response relationships between energy availability and bone turnover in young exercising women. J Bone Miner Res. 2004 Aug;19(8):1231-40. doi: 10.1359/JBMR.040410. Epub 2004 Apr 19. PMID 15231009